CLINICAL TRIAL: NCT00520832
Title: A Pilot Study Of The Effects Of Microcurrent On Three Sleep Surveys
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SR0524070091
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Primary Insomnia
Keywords: Primary Insomnia; Microcurrent Therapy; Sleep Surveys
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MC-E (Experimental): 20 minutes of sub-threshold microcurrent 2 hours before bedtime per day for 21 days.
  Interventions: Device: Microcurrent
- MC-P (Placebo Comparator): Participants will receive a device identical to the active device used in the experimental condition, but which produces no current.
  Interventions: Device: Microcurrent

INTERVENTIONS:
Device: Microcurrent — 20 minutes of sub-threshold microcurrent 2 hours before bedtime per day for 21 days.
  Arms: MC-E
Device: Microcurrent — Participants will receive a device identical to the active device used in the experimental condition, but which produces no current.
  Arms: MC-P

SUMMARY:
Participants identified as having primary insomnia will be randomly assigned to groups receiving microcurrent stimulation or sham in a double-blind randomized controlled trial. The microcurrent device used is FDA approved for the treatment of insomnia.

The hypothesis is that the experimental group will have significantly improved scores on three sleep surveys after treatment while the sham group will not.

ELIGIBILITY:
Inclusion Criteria:

* Student, Faculty or Staff
* Age 18 - 40
* Symptoms of primary insomnia

Exclusion Criteria:

* No implanted electric devices
* No local infection, injury or malignancy
* No history of seizure or other neurological disorders
* No current use of prescription or other substances that could effect sleep quality or quantity
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI)
Epworth Sleepiness Scale
Insomnia Severity Index

CONTACTS AND LOCATIONS:
Overall Officials: Rodger Tepe, PhD, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States